CLINICAL TRIAL: NCT05003154
Title: Comparison of Conventional Mode and Combined Digitalized Mode of Management for Gestational Diabetes Mellitus in China
Brief Title: Digitalized Management Exploration for Gestational Diabetes Mellitus in China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Hangzhou Jianhai Technology Company Limited (Unknown); Quzhou Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDMDM2021
Record Dates: First submitted 2021-07-30; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional management group (No Intervention): Received conventional management based on Guidelines for GDM in China
- Digitalized management group (Experimental): Reveived conventional management and digitalized management
  Interventions: Other: Digitalized management

INTERVENTIONS:
Other: Digitalized management — In addition to conventional management, Patients also receive digitalized management, which provides personalized guidance in diet, excercise, prenatal visit, blood glucose monitoring,etc., from artificail intelliegence (AI) supevised by obstetricians, through a smartphone application and some werable devices (like sports bracelet).
  The pivotal AI are based on clinical experience from obstetricians, therapeutic principle from official Guidelines and abundant data in previous work, and it will works under strict supervision.
  Arms: Digitalized management group

SUMMARY:
Gestational diabetes mellitus (GDM) can lead to adverse perinatal and long-term outcomes, and it is so important to manage this disease in pregnancy. Digitalized managements have been proved economical and effective in some chronic diseases like type II diabetes mellitus. The purpose of the current study was to develop and evaluate a digitalized mode for GDM management using mobile healthcare and some wearable devices. Subjects were randomly divided into a conventional management group and combined digitalized management group after diagnosed with GDM during 24-28 weeks of gestation. The conventional mangement group received conventional GDM management and could freely use the mobile healthcare application. The mobile management group received digitalized healthcare services from artificial intelligence under the supervision of obstetricians, in addition to conventional management. The effectiveness of digitalized management were evaluated mainly through the result values of the labotatory tests related to blood glucose controlling and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. The age of 18-45 years, single pregnancy, Han nationality;
2. GDM diagnosed between 24 to 28 weeks of gestation, either of the following: fasting plasma glucose ≥5.1 mmol/L, 60-minute plasma glucose ≥10.0 mmol/L, 120-minute plasma glucose ≥8.5 mmol/L, during a 75g oral glucose tolerance test (OGTT).
3. Plan to deliver the baby in Women's Hospital School Of Medicine Zhejiang University;
4. Can operate mobile phones and related software;
5. Voluntary participation in this study;
6. Education background: junior high school or above.

Exclusion Criteria:

1. Type I or II or other non GDM diabetes mellitus;
2. Severe pregnancy complications or complications: such as malignant tumor, preeclampsia, severe intrahepatic cholestasis of pregnancy syndrome, pregnancy with antiphospholipid antibody syndrome, severe anemia (hemoglobin<90g/L, etc.), cardiac insufficiency cardiovascular disease (such as myocardial infarction, heart failure, pulmonary hypertension, stroke history, coronary heart disease, valvular heart disease, etc.), stroke (moderate), liver disease (such as hepatic insufficiency, acute viral hepatitis, etc.), lung disease (such as restrictive lung disease, emphysema, liver cirrhosis, pulmonary heart disease, etc.), kidney disease (such as nephrotic syndrome, chronic nephritis, renal insufficiency, etc.), chronic hypertension, thyroid disease (such as hyperthyroidism, hypothyroidism, thyroiditis, etc.), other endocrine diseases (such as Cushing's syndrome Acromegaly, venous or arterial thromboembolic diseases, rheumatic immune diseases, etc;
3. The combined conditions that may affect the diet exercise therapy include severe food allergy, dyskinesia (physical disability), history of bariatric surgery, major gastrointestinal diseases (such as gastrointestinal bleeding, inflammatory bowel disease, gastrointestinal tumor, active stage of peptic ulcer, chronic intestinal obstruction, etc.), restrictive lung disease, history of two or more adverse abortions, placenta previa, repeated and persistent bleeding threatened abortion, threatened premature birth, hyperemesis gravidarum, vegetarians, etc;
4. Other conditions: such as mental disorders, cervical incompetence, genital tract deformity, etc;
5. Patients who are taking medicine that may affect glucose metabolism, such as ritodrine, prednisone, etc;
6. Patients who are participating in other clinical studies;
7. The researchers believe patients who are not suitable for this study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Concentration of glycosylated hemoglobin A1c | 37-42 weeks of gestation
  Reflecting the average glucose level in the last 8-12 weeks

SECONDARY OUTCOMES:
Rate of neonate large for gestational age | At the 1 day of delivery
  May reflecting maternal glucose level in pregnancy
rate of caesarean as the delivery mode | At the 1 day of delivery
  An indicator associated with fetal weight or perinatal condition
Hospitalization cost of neonate and puerperae for delivery | At the 1 day discharging from hospital
  A health economic indicator
Proportion of patients with abnormal resulets of postnatal oral glucose tolerance test | 42 days postpartum
  Reflecting postpartum glucose metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Danqing Chen, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Du M, Yi S, Wei Y, Jiang Y, Bao S, Lu J, Chen D. Effect of FSL-CGM on Maternal and Neonatal Outcomes in GDM: A Propensity Score Matching Study in Hangzhou, China. Diabetes Ther. 2025 Jul;16(7):1385-1397. doi: 10.1007/s13300-025-01749-0. Epub 2025 May 12. PMID 40353986